CLINICAL TRIAL: NCT06233305
Title: Effect of Physical Therapy and/or Platelet Rich Plasma Injection in People With Knee Cruciate Ligament Injuries: an Observative Study
Brief Title: Effect of Physical Therapy and/or Platelet Rich Plasma Injection in People With Knee Cruciate Ligament Injuries
Status: Recruiting | Type: Observational
Sponsor: Taipei Hospital, Ministry of Health and Welfare (Other)
Responsible Party: Sponsor
Other Study IDs: 202414
Record Dates: First submitted 2024-01-22; First posted 2024-01-31 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Anterior Cruciate Ligament Tear; Posterior Cruciate Ligament Tear
Keywords: PRP; Therapeutic exercise; Modality physical therapy
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background:

The anterior cruciate ligament(ACL) , one of the major ligaments in the knee joint which connects the posterior aspect of the lateral femoral condyle to the anterior intercondylar area of the tibia. It plays a crucial role in maintaining knee joint stability, preventing excessive rotation of the tibia, and controlling the angles of knee valgus and varus. Additionally, the ACL contains mechanoreceptors that contribute to proprioception input. Acute ACL injuries are characterized by joint effusion, instability, and reduced range of motion. In the chronic phase, instability and pain may occur during rotational and cutting movements.

Currently, regenerative injection therapies such as high-concentration platelet-rich plasma (PRP)and bone marrow concentrate (BMC) are being explored for ACL repair. Studies have found that postoperative administration of high-concentration PRP significantly reduces pain and improves knee joint function for a duration of 3 to 6 months, but these effects are not sustained beyond 12 months. In addition, some research indicates that high-concentration PRP does not enhance graft healing or improve knee joint stability.

Method:

This is a single-institution, single-blind, observational study conducted by the rehabilitation department of a public hospital. The study aims to recruit 40 participants with anterior cruciate ligament (ACL) or posterior cruciate ligament (PCL) injuries. The treatment intervention is collaboratively determined by the physician and the participant during the clinic visit. Subsequently, a therapist, unaware of the treatment details, conducts baseline assessments, including basic information collection, balance testing, gait analysis, timed up and go test, muscle strength evaluation, and subjective knee assessment questionnaire. Additionally, a physician, blinded to the treatment content, employs ultrasound to assess ligament elasticity. Follow-up assessments are conducted for the same parameters two months later.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 to 80 years old.
2. Magnetic Resonance Imaging (MRI) shows partial tearing of the anterior cruciate ligament (ACL) or posterior cruciate ligament (PCL), possibly combined with injuries to the medial collateral ligament (MCL) or meniscus.
3. No surgical treatment has been undergone.

Exclusion Criteria:

1. Had knee joint diseases or undergone knee joint surgery before the injury.
2. Surgical intervention is required for severe damage to knee joint ligaments, meniscus, or articular tissues, such as complete rupture of lateral ligaments or full-thickness cartilage injuries.
3. Suffers from diseases affecting physical activity function, such as stroke or nerve damage.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study subjects were sampled from the Rehabilitation Department of the Taipei Hospital, Ministry of Health and Welfare, with an anticipated enrollment of 40 individuals with anterior cruciate ligament (ACL) knee injuries
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-01-03 (Actual); Primary Completion 2024-12-27 (Estimated); Study Completion 2025-03-27 (Estimated)

PRIMARY OUTCOMES:
Balance Sensing Test | Pre-treatment assessment, approximately one month later perform a mid-term assessment, and two months later, conduct a post-treatment assessment.
  Subjects were instructed to wear knee protectors(KNEESUP Care ) equipped with 3D gyroscopes which made from Conzion and subjects were asked to perform three trials of open-eye single-leg standing and three trials of closed-eye single-leg standing. The dynamic sensing system software recorded the time spent in single-leg standing and analyzed parameters such as balance area, anterior-posterior and medial-lateral displacement of the knee joint, and differences between the two feet.
Gait Analysis | Pre-treatment assessment, approximately one month later perform a mid-term assessment, and two months later, conduct a post-treatment assessment.
  Subjects were instructed to wear knee protectors(KNEESUP Care ) equipped with 3D gyroscopes which made from Conzion. Gait analysis involves having the subjects walk back and forth for six meters while wearing the device, with the software analyzing differences in the gait of both feet.
Time up and go test | Pre-treatment assessment, approximately one month later perform a mid-term assessment, and two months later, conduct a post-treatment assessment.
  Subjects were instructed to wear knee protectors(KNEESUP Care ) equipped with 3D gyroscopes which made from Conzion. The patient stand up from the chair, walking three meters forward, turn around, and return to the chair to sit down.The KNEESUP will calculate the total time needed
Muscle Strength Test | Pre-treatment assessment, approximately one month later perform a mid-term assessment, and two months later, conduct a post-treatment assessment.
  Quantify muscle strength of knee extensors and knee flexors using a hand-held dynamometer(ISOFROCE GT-300) which made from OG WELLNESS
International Knee Documentation Committee | Pre-treatment assessment, approximately one month later perform a mid-term assessment, and two months later, conduct a post-treatment assessment.
  A total of 18 items were assessed, covering aspects such as symptoms, physical activity, and functionality. Each item was scored on a sequential scale, with higher scores indicating lower symptoms and higher functionality. The sum of all scores was calculated and then converted into a scale ranging from 0 to 100.
Ligament elasticity | Pre-treatment assessment, approximately one month later perform a mid-term assessment, and two months later, conduct a post-treatment assessment.
  Utilizing shear wave elastography, elastic images are generated by inducing shear waves within the tissue using acoustic pressure waves. The propagation speed of these waves is directly proportional to the square root of the tissue's elastic modulus. The elasticity coefficient of the anterior cruciate ligament is measured in patients at various degrees of knee flexion.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Hospital, Ministry of Health and Welfare, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No